CLINICAL TRIAL: NCT06042595
Title: Predicting Premature Treatment Termination in Inpatient Psychotherapy: A Machine Learning Approach
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Simone Jennissen, Principal Investigator, University Hospital Heidelberg
Other Study IDs: Dropout-Prediction-2023
Record Dates: First submitted 2023-08-11; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Premature Treatment Termination; Dropout Prediction; Inpatient Psychotherapy; Machine Learning
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Psychotherapy — Patients treated at the inpatient psychotherapy unit of the University Hospital receive 8 to 10 weeks of multimodal psychotherapeutic treatment. Treatment consists of individual as well as group psychodynamic therapy. Additionally, patients receive an individual combination of music, art, relaxation and body-oriented group therapy. Therapeutic treatment is provided by a multiprofessional, interdisciplinary team of psychotherapists with either a medical or psychology degree, art and music therapists, specialist nurses, social workers, and physiotherapists.

SUMMARY:
The study aims to develop a prediction model of premature treatment termination in psychosomatic hospitals using a machine learning approach.

DETAILED DESCRIPTION:
The aim of the study is to identify risk factors that lead to or predict premature treatment termination in psychosomatic hospitals. In the long-term, the study shall help to develop more precise prediction models that can enhance communication between therapists and patients about potential dropout and- if necessary- adaption of treatment in using a feedback loop.

Since it is still not clear which variables play a major role in predicting treatment termination in psychosomatic hospitals, the study design is exploratory and includes a broad range of intake patient characteristics. The purpose of this study is hereby, to develop a prediction model based on the information that are routinely assessed at intake. Therefore, three kind of variables are planned to be included: (1) demographic and other clinical variables (e.g. age, gender, ICD-10 diagnoses), (2) psychological questionnaire data (e.g. PHQ, SF-12, EB-45, IIP-32, OPD-SFK), and (3) physiological data (e.g. routine laboratory data, blood pressure). For the study, all patients that started inpatient psychotherapy at the medical centre Heidelberg between 2015 and January 2022 will be included, resulting in a sample size of approximately N = 2000. As the average dropout rate based on meta analytical results is around 20%, one can assume that up to 400 patients prematurely dropped out of treatment.

To calculate the prediction model, it is planned to use a machine learning approach which is highly functional in big data sets. Using a Random Forest Model for binary outcomes (regular treatment length vs. premature treatment termination) it is envisioned to identify variables that contribute to the prediction of premature treatment termination at intake. Additionally, waiting list effects will be considered by taking into account the waiting duration between the initial intake interview and the moment of the hospital admission. Therefore, the study will, for the first time, investigate a prediction model for premature treatment termination in inpatient psychotherapy including clinically relevant physiological data as well as waiting time effects in preparation of the psychosomatic treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients of at least 18 years of age
* included in inpatient psychotherapy treatment program in a hospital for psychosomatic medicine
* provided information about admission and discharge date

Exclusion Criteria:

* bipolar, acute psychotic or substance abuse disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients being treated at the inpatient unit of University Hospital Heidelberg, department for psychosomatic medicine.
Sampling Method: Non-Probability Sample
Enrollment: 2023 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Premature treatment termination (vs. treatment completion) | Premature treatment termination will be operationalized as a dummy variable. Regular treatment duration is 8 weeks of inpatient psychotherapy. Data will be reported for 7 years of continuous study enrolment (01/2015 - 01/2022).
  Premature treatment termination will be classified based on the treatment duration. Classification will be made retrospectively for each patient based on the duration of the inpatient treatment and if applicable (duration < 49 days) on the hospital discharge letter to screen for reasons of the shorter treatment duration.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Dinger-Ehrenthal, Prof. Dr., Study Director — Department of Psychosomatic Medicine and Psychotherapy, Medical Faculty, Heinrich-Heine University Düsseldorf

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because study data is provided by mental health patients and is therefore subject to strict protection.